CLINICAL TRIAL: NCT03968042
Title: Efficacy and Safety of Nerve Growth Factor or Edaravone on Alcohol-induced Brain Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Peng, Professor, Director of Department of Neurology, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-13-NGF-EDV
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Alcohol-induced Brain Injury
Keywords: Alcohol-induced brain injury, atrophy, demyelination
MeSH Terms: conditions — Atrophy; Demyelinating Diseases | interventions — Nerve Growth Factor; Edaravone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular treatment (RT) (Placebo Comparator): Combination of vitamin B1, B6, C, E and mecobalamine
  Interventions: Drug: Combination of vitamin B1, B6, C, E and mecobalamine
- RT with NGF (Experimental): Nerve growth factor adding to regular treatment
  Interventions: Drug: Nerve Growth Factor; Drug: Combination of vitamin B1, B6, C, E and mecobalamine
- RT with EDV (Experimental): Edaravone adding to regular treatment
  Interventions: Drug: Edaravone; Drug: Combination of vitamin B1, B6, C, E and mecobalamine

INTERVENTIONS:
Drug: Nerve Growth Factor — Intramuscular injection for 2 weeks
  Arms: RT with NGF
Drug: Edaravone — Intravenous injection for 2 weeks
  Arms: RT with EDV
Drug: Combination of vitamin B1, B6, C, E and mecobalamine — Medications of combination of vitamin B1, B6, C, E and mecobalamine for 6 months

SUMMARY:
Alcohol is one of most common harmful substance, and alcohol intake brings great burden on health worldwide. Excess alcohol intake may lead to alcohol-related brain injuries and cognitive impairment. Although both nerve growth factor and antioxidative treatment were effective to relieve alcohol-related injuries in central nervous system in the preclinical studies, there is no relevant clinical trial about their efficacy and safety on patients. Since nerve growth factor and one of the antioxidative medication, edaravone, have been used in some neural diseases in clinical trials, we tend to evaluate the efficacy and safety of nerve growth factor, or edaravone on alcohol-induced brain injuries. The study is a randomized-controlled study and the patients will be assigned into one of the following three groups randomly: (1) regular treatment (combination of vitamin B1, B6, C, E and mecobalamine) with nerve growth factor for 2 weeks and subsequently regular treatment for 6 months; (2) regular treatment (RT) with edaravone for 2 weeks and subsequently RT for 6 months; (3) RT alone for 6 months. The patients will be followed up for 6 months. Cognitive functions, recurrence of alcohol dependence, duration of abstention, alcohol intake, craving for alcohol and other psychological assessments will be recorded and compared among the 3 treatment groups and the efficacy of nerve growth factor or edaravone will be evaluated in our study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as alcohol dependence according to DSM-IV criteria
* MRI-proved demyelinating lesions or atrophy in the brain of the patient
* No definite history of neurological diseases and psychological problems
* Volunteer to participate the study, cooperate to be followed up

Exclusion Criteria:

* Acute withdrawal state and CIWA score > 9
* With other neurological diseases and psychological problems
* With ever brain trauma and damage
* With other psychological medications or other substance dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive improvement | 2 weeks
  Executive function by digit symbol substitute test (DSST) ranging from 0 to 90. Higher score indicates better executive function.
Cognitive improvement | 2 months
  Executive function by digit symbol substitute test (DSST) ranging from 0 to 90. Higher score indicates better executive function.
Cognitive improvement | 3 months
  Executive function by digit symbol substitute test (DSST) ranging from 0 to 90. Higher score indicates better executive function.
Cognitive improvement | 6 months
  Executive function by digit symbol substitute test (DSST) ranging from 0 to 90. Higher score indicates better executive function.
Cognitive assessment | 3 months
  Cognitive assessment by Montreal Cognitive Assessment (MoCA) ranging from 0 to 30. Lower score indicates worse cognitive function.
Cognitive assessment | 6 months
  Cognitive assessment by Montreal Cognitive Assessment (MoCA) ranging from 0 to 30. Lower score indicates worse cognitive function.

SECONDARY OUTCOMES:
The rate of relapse of alcohol dependence after discharge from hospital | 2 months
  Recurrence of alcohol dependence
Duration of abstinence | 6 months
  The total time or period without any intake of alcohol during follow ups
Alcohol intake | 2 weeks, 2 months, 3 months, 6 months
  Diaries of alcohol intake in different time of the follow ups
Craving for alcohol | 2 weeks, 2 months, 3 months, 6 months
  Craving assessment for alcohol by Obsessive Compulsive Drinking Scale (OCDS) ranging from 0 to 40. Higher score of OCDS indicates more desire for alcohol.
Psychological assessment - Anxiety | 2 weeks, 2 months, 3 months, 6 months
  Psychological assessment by Generalized Anxiety Disorder-7 (GAD-7) ranging from 0 to 21. Higher score indicates more severer anxiety.
Psychological assessment - Depression | 2 weeks, 2 months, 3 months, 6 months
  Psychological assessment by Patient Health Questionnaire-9 (PHQ-9) ranging from 0 to 27. Higher score indicates more severer depression.
Psychological assessment - Sleep | 2 weeks, 2 months, 3 months, 6 months
  Psychological assessment by Pittsburgh Sleep Quality Index (PSQI) ranging from 0 to 21. Higher score indicates worse sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun YY, Li Y, Wali B, Li Y, Lee J, Heinmiller A, Abe K, Stein DG, Mao H, Sayeed I, Kuan CY. Prophylactic Edaravone Prevents Transient Hypoxic-Ischemic Brain Injury: Implications for Perioperative Neuroprotection. Stroke. 2015 Jul;46(7):1947-55. doi: 10.1161/STROKEAHA.115.009162. Epub 2015 Jun 9. PMID 26060244
- [Background] Kaste M, Murayama S, Ford GA, Dippel DW, Walters MR, Tatlisumak T; MCI-186 study group. Safety, tolerability and pharmacokinetics of MCI-186 in patients with acute ischemic stroke: new formulation and dosing regimen. Cerebrovasc Dis. 2013;36(3):196-204. doi: 10.1159/000353680. Epub 2013 Oct 12. PMID 24135530
- [Background] Munakata A, Ohkuma H, Nakano T, Shimamura N, Asano K, Naraoka M. Effect of a free radical scavenger, edaravone, in the treatment of patients with aneurysmal subarachnoid hemorrhage. Neurosurgery. 2009 Mar;64(3):423-8; discussion 428-9. doi: 10.1227/01.NEU.0000338067.83059.EB. PMID 19240603
- [Background] Writing Group; Edaravone (MCI-186) ALS 19 Study Group. Safety and efficacy of edaravone in well defined patients with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2017 Jul;16(7):505-512. doi: 10.1016/S1474-4422(17)30115-1. Epub 2017 May 15. PMID 28522181
- [Background] Apfel SC, Kessler JA, Adornato BT, Litchy WJ, Sanders C, Rask CA. Recombinant human nerve growth factor in the treatment of diabetic polyneuropathy. NGF Study Group. Neurology. 1998 Sep;51(3):695-702. doi: 10.1212/wnl.51.3.695. PMID 9748012
- [Background] Riggs JE. Recombinant human nerve growth factor in the treatment of diabetic polyneuropathy. Neurology. 1999 Apr 22;52(7):1517-8. doi: 10.1212/wnl.52.7.1517-a. No abstract available. PMID 10227655
- [Background] McArthur JC, Yiannoutsos C, Simpson DM, Adornato BT, Singer EJ, Hollander H, Marra C, Rubin M, Cohen BA, Tucker T, Navia BA, Schifitto G, Katzenstein D, Rask C, Zaborski L, Smith ME, Shriver S, Millar L, Clifford DB, Karalnik IJ. A phase II trial of nerve growth factor for sensory neuropathy associated with HIV infection. AIDS Clinical Trials Group Team 291. Neurology. 2000 Mar 14;54(5):1080-8. doi: 10.1212/wnl.54.5.1080. PMID 10720278
- [Background] Lambiase A, Rama P, Bonini S, Caprioglio G, Aloe L. Topical treatment with nerve growth factor for corneal neurotrophic ulcers. N Engl J Med. 1998 Apr 23;338(17):1174-80. doi: 10.1056/NEJM199804233381702. PMID 9554857
- [Background] Petty BG, Cornblath DR, Adornato BT, Chaudhry V, Flexner C, Wachsman M, Sinicropi D, Burton LE, Peroutka SJ. The effect of systemically administered recombinant human nerve growth factor in healthy human subjects. Ann Neurol. 1994 Aug;36(2):244-6. doi: 10.1002/ana.410360221. PMID 8053664
- [Background] Zhou F, Wu P, Wang L, Wang HT, Zhang SB, Lin Y, Zhong H, Chen YH. The NGF point-injection for treatment of the sound-perceiving nerve deafness and tinnitus in 68 cases. J Tradit Chin Med. 2009 Mar;29(1):39-42. doi: 10.1016/s0254-6272(09)60029-7. PMID 19514187
- [Background] Wu ZH, Huang J, Gao WH, Wang AL, Jia Q, Chen B, Xu S, Gu YH. [Effect of nerve growth factor on the promotion of sensory recovery of large skin graft in patients]. Zhonghua Shao Shang Za Zhi. 2007 Dec;23(6):440-3. Chinese. PMID 18457257
- [Derived] Wang H, Liu L, Zhou X, Guan Y, Li Y, Chen P, Duan R, Yang W, Rong X, Wu C, Yang J, Yang M, Jia Y, Hu J, Zhu X, Peng Y. Efficacy and safety of short-term edaravone or nerve growth factor add-on therapy for alcohol-related brain damage: A multi-centre randomised control trial. Addiction. 2024 Apr;119(4):717-729. doi: 10.1111/add.16398. Epub 2023 Dec 4. PMID 38049955